CLINICAL TRIAL: NCT03783247
Title: Pericapsular Nerve Group Block Versus Fascia Iliaca Block for Hip Arthroplasty: a Randomized Controlled Trial
Brief Title: Peri-capsular Nerve Group Block Versus Fascia Iliaca Block for Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan Mohamed Ali, associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Swelam PENG block
Record Dates: First submitted 2018-12-18; First posted 2018-12-21 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Post Operative Pain Management

STUDY DESIGN:
Intervention Model Description: randomized double-blinded
Who Masked: Participant, Outcomes Assessor
Masking Description: To achieve double blinding, patients will receive the block by the anesthetist. Another doctor not involved in the block procedure will evaluate the patients postoperatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIB (Experimental): hip fracture with fascia Iliaca block
  Interventions: Procedure: Fascia Iliaca BLock
- PENG (Experimental): Hip fracture with Pericapsular nerve group block
  Interventions: Procedure: Pericapsular nerve group block

INTERVENTIONS:
Procedure: Pericapsular nerve group block — The regional block was performed with the patient in the supine position. A curvilinear low-frequency ultrasound probe (2-5MHz) was initially placed in a transverse plane over the AIIS and then aligned with the pubic ramus by rotating the probe counterclockwise approximately 45 degrees (Figs. 2, 3). In this view, the IPE, the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle were observed. A 22-gauge, 80-mm needle was inserted from lateral to medial in an in-plane approach to place the tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. Following negative aspiration, the local anesthetic solution (20ml of bupivacaine 0.25%) was injected in 5-mL increments while observing for adequate fluid spread in this plane for a total volume of 30 mL
  Other Names: PENG
  Arms: PENG
Procedure: Fascia Iliaca BLock — In supine position, a high frequency linear probe will be placed in the inguinal crease. Scan starting laterally from the femoral artery and nerve in inguinal crease to identify the sartorius muscle, tracing the muscle until it's origin to anterior superior iliac spine. The shadow of the bony of iliac crest & iliacus muscle will be seen, the end point of the injection is deep to the fascia iliaca and above the iliacus muscle in the lateral part of the iliacus muscle. After negative aspiration, 30 mL of 0.25 % of bupivacaine will be injected under the fascial plane incrementally, aspirating every 5 ml.
  Other Names: FIB
  Arms: FIB

SUMMARY:
In this study, the investigator will examine the efficacy of Pericapsular nerve group (PENG) block in hip surgeries as a post-operative pain management technique in comparison with fascia Iliaca block in hip surgeries

DETAILED DESCRIPTION:
Hip fracture is a common orthopedic emergency in the elderly, and it is associated with significant morbidity and mortality.1 Surgical reduction and fixation are the definitive treatment in most patients.2 Effective perioperative analgesia that minimizes the need for opioids and related adverse effects (such as delirium) is essential in this patient population.

Regional analgesic techniques, including femoral nerve (FN) block, fascia iliaca block (FIB), and 3-in-1 FN block, are popular analgesic strategies, due mainly to their opioid-sparing effects and reduction in opioid-related adverse effects. The effect size of analgesia from these blocks is only moderate, and literature suggests that the obturator nerve (ON) is not covered.

The anterior hip capsule is innervated by the ON, accessory obturator nerve (AON), and FN as reported by previous anatomic studies. The anterior capsule is the most richly innervated section of the joint, suggesting these nerves should be the main targets for hip analgesia. A recent anatomical study by Short et al15 confirmed the innervation of the anterior hip by these 3 main nerves but also found that the AON and FN play a greater role in the anterior hip innervation than previously reported. This study also identified the relevant landmarks for those articular branches. The high articular branches from FN and AON are consistently found between the anterior inferior iliac spines (AIIS) and the iliopubic eminence (IPE), whereas the ON , close to the inferomedial acetabulum. Using this information, the investigator developed an ultrasound-guided technique for blockade of these articular branches to the hip, the PENG (PEricapsular Nerve Group) block. In this study, the investigator will examine the efficacy of PENG block in hip surgeries as a post-operative pain management technique in comparison with fascia Iliaca block in hip surgeries

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for hip replacement surgeries e.g. hip hemiarthroplasty, total hip arthroplasty under subarachnoid block (SAB)

Exclusion Criteria:

* Coagulopathy
* infection at the injection site
* allergy to local anesthetics
* severe cardiopulmonary disease (≥ASA IV)
* diabetic or other neuropathies
* patients receiving opioids for chronic analgesic therapy
* contraindication to spinal anesthesia
* inability to comprehend visual analog scale (VAS).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-15 (Estimated); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-06-20 (Estimated)

PRIMARY OUTCOMES:
morphine consumption | 24 hours
  total morphine consumption over 24 hours

SECONDARY OUTCOMES:
pain scale Visual analogue Scale | 24hours
  Using a ruler, the score is determined by mea-suring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
muscle power | 24 HOURS
  Assessment of quadriceps femoris muscle strength: For motor block assessment, the patient will be in supine position and the patient's knee will be fully flexed, and the patient will be asked to extend it. The motor block is classified as follows: grade 0; normal muscle power, grade I; motor weakness, grade II; complete motor paralysis

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided